CLINICAL TRIAL: NCT02814981
Title: Hydroxyzine and Risk of Prolongation of QT Interval
Acronym: HYDROXYZINE-QT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A15-D44-VOL.27
Record Dates: First submitted 2016-06-17; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Hydroxyzine; Long QT Syndrome
Keywords: hydroxyzine; Long QT
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
On 04/30/2015, ANSM (the National Security Agency of Medicines and Health Products) shared an information for general practicioners, pediatricians, anesthesiologists, dermatologists, geriatricians, psychiatrists, community pharmacists and hospital about using hydroxyzine and the associated risk of QT prolongation on the electrocardiogram.

Drugs containing hydroxyzine (the best known and most used is the Atarax®) are used in France in various indications including the treatment of minor manifestations of anxiety, premedication with general anesthesia and the symptomatic treatment of urticaria.

A prolonged QT interval is a known risk factor for occurrence of torsades de pointes which can cause sudden death. We distinguish congenital and acquired long QT interval. The main cause of acquired long QT interval is a drug inhibition of the HERG potassium channel 1. Many drugs have been reported to cause sudden death by prolongation of QT interval and occurrence of torsades de pointes (macrolides, anti -arythmics, some psychotropic ...) The molecules based on hydroxyzine are known to be at risk of prolongation of QT interval in an experimental point of view but is not clearly identified in daily clinical practice. Pharmacology unit of Caen was the first to publish a case of QT prolongation under hydroxyzine . Through this publication, associated with other clinical data, hydroxyzine has been added to the list of drugs that can induce QT prolongation .

Despite these recent recommendations, it does not seem that hydroxyzine prescriptions were changed daily and therefore the risk of QT prolongation persists. We therefore propose the study of the impact of hydroxyzine on the QT interval measured on the electrocardiogram in patients hospitalized at the University Hospital of Caen.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at the University Hospital of Caen with a new prescription of oral hydroxyzine by their referring doctor.
* Patient 'stable' in hospital in a health service or surgery.
* Age > 18 years old.

Exclusion Criteria:

* Unstable Patient hospitalized in an intensive care unit or intensive care.
* Patient refusing participation in the study.
* Age <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients hospitalized in Caen University Hospital with a prescription of hydroxyzine drug.
  From there, after informing the patient, we will collect the measurement of QT interval before introducing hydroxyzine and the same measure will be performed again on the 3rd day.
  QT will be corrected by heart rate by Bazett's formula (the most commonly used) and Fridericcia (most reliable). Reproducibility of analyzes inter and intra-individual will be carried out to ensure the reliability of the measurements.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Measure of the corrected QT interval in ms | 1 day
  Measure of corrected QT interval with Bazett and Frediriccia method , in DII and V5.

SECONDARY OUTCOMES:
Number of Incoming of torsade de pointe | up to 1 month
  polymorphic ventricular tachycardia with a characteristic illusion of a twisting of the QRS complex
risk of sudden death by ventricular arythmia | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: Yes